CLINICAL TRIAL: NCT06991816
Title: The Brain&Senses Study Impact of Multi Sensory Impairments on the Progression of Cognitive Decline and Reduction of Quality of Life in People Over 50ies
Brief Title: The Brain&Senses Study
Status: Not yet recruiting | Type: Observational
Sponsor: University of Campania Luigi Vanvitelli (Other)
Collaborators: Ospedali Riuniti Marche Nord, Fano-Pesaro Hospital (Unknown)
Responsible Party: Principal Investigator, Arianna Di Stadio, Associate Professor of Otolaryngology, University of Campania Luigi Vanvitelli
Other Study IDs: NAFA2025
Record Dates: First submitted 2025-03-24; First posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease; Parkinson
Keywords: Cognitive Decline; Smell Loss; Vertigo/ Dizziness; Hearing Loss
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Anosmia; Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this longitudinal observational study is to evaluate the impact of sensory deficits (smell, hearing and balance on cognitive decline and quality of life in the medium term (5 years)) on a population of patients over 55.

Patients will be evaluated by a neurologist, a neuropsychologist and an otolaryngologist who will perform olfactory, auditory and vestibular tests.

The acquired data will then be analyzed with multivariate analysis to understand the effect of multisensory deficit on both cognition and quality of life with a particular focus on depression.

The primary objective will be the evaluation of multiple deficits on cognition, the secondary will be aimed at understanding whether one sensory deficit more than another, e.g. smell versus hearing, will have a greater impact on the patient's conditions.

DETAILED DESCRIPTION:
Evaluation protocol

Enrollment phase: the subjects will be recruited through recruitment at the Department of Neurology of the Fano hospital and the various associations supporting patients with cognitive impairment in the area. The subjects who meet the inclusion and exclusion criteria for the cohort will be contacted and invited for the ENT evaluations that will be carried out in the Department of Otolaryngology of the FANO hospital.

Inclusion criteria: patients between 60 and 85 years of age, in general good health, in the absence of known severe psychiatric disorders, available to be included in the study and to follow the 5-year follow-up.

Exclusion criteria: Obstructive nasal problems, Previous endoscopic nose + paranasal sinus surgery, Chronic use of cortisone spray and/or systemic, Subjects with previous stroke and outcomes, Subjects with history of stroke in the last 3 years without outcomes, Head trauma in the last 24 months, Previous ear surgery, Patients who have been exposed to chemical agents without protection for work, e.g. carpenters and previous Covid with outcomes (olfactory, vestibular, auditory and cognitive "brain fog")

Neurology

Total evaluation time 20-30 minutes

All patients will be clinically evaluated in neurology; specifically, vertical gaze and archaic reflexes (muzzle and palm-chin) will be evaluated. From a laboratory point of view, blood count with formula, AST, ALT, Sodium and Potassium, creatinine, TSH, dosage of Vitamin B12 and folates will be performed.

NeuroPsychology

Total evaluation time 35-65 minutes

Patients will be subjected to the standard battery of neuropsychological tests which includes the MMSE, MoCA, working and short memory tests.

The duration of the psychological tests may vary based on the patient's conditions.

NEUROPSYCHOLOGICAL BATTERY The subjects of the study were administered a neuropsychological battery consisting of the following tests

Mini Mental State Examination (MMSE) (Folstein et al., 1975; Magni et al., 1996): is an 11-item screening test that assesses the level of basic cognitive functioning. This test consists of 11 domains that assess:

* Temporal Orientation;
* Spatial Orientation;
* Mnemonic Recall of 3 items;
* Attention and Calculation;
* Recall of the 3 items mentioned in the previous exercise;
* Language and Practice. The test score ranges from 0 to 30 and the points obtained in each item are added together. The raw score obtained is corrected for the participant's level of education and age.

Montreal Cognitive Assessment (MoCA) (Nasreddine et al., 2005; Conti et al., 2015): This is a test consisting of several trials with a total of 30 items. The short-term memory task (5 items) consists of two learning trials with five names and a delayed recall after about 5 minutes. Visual-spatial ability is assessed with a clock drawing task (3 points) and a copy of a three-dimensional cube (1 point). Several aspects of executive function are assessed with a Trail Making B task (1 point), a phonemic fluency task (1 point) and a two-item verbal abstraction task (2 points). Attention, concentration and working memory are assessed with a sustained attention task (target identification by typing; 1 point), a serial subtraction task (3 points) and a forward and backward digit task (1 point each). Language is assessed using a three-item naming task with unfamiliar animals (lion, camel, rhinoceros; 3 points), the repetition of two words (2 points), the repetition of two syntactically complex sentences (2 points) and the above-mentioned fluency task. Finally, time and place orientation is assessed (6 points). The test score ranges from 0 to 30 and the points obtained in each item are added together. The raw score obtained is corrected for the participant's level of education and age.

Frontal Assessment Battery (FAB) (Dubois et al., 2000; Apollonio et al., 2005): is a screening battery designed to assess global executive functioning. It consists of 6 cognitive and behavioural tests, each of which has a score ranging from 0 to 3 (range 0-18):

* Conceptualisation of similarity: the subject is asked to identify the relationship between three stimuli (e.g. "How are a rose, a daisy and a tulip similar?");
* Phonemic fluency;
* Motor programming (Luria series): the subject has to reproduce the motor series (punching, cutting, flattening) performed by the examiner;
* Response to conflicting instructions: the subject has to carry out a series of exercises several times, together with the examiner, according to the instructions given by the examiner ("Knock twice if I knock once"; "Knock once if I knock twice"). This is a very good test for assessing attention and interference sensitivity;
* Go-no-go task: same principle as the previous test, but in this case the instructions given are more useful for assessing inhibitory control capacity ("Knock once if I knock once"; "Don't knock if I knock twice");
* Prehension behaviour: the subject is asked to place their hands in a "clamshell" position (resting on a surface, palms up). Then, without saying anything, the examiner brings his hands close to those of the respondent and touches their palms. The aim of the exercise is to assess environmental autonomy by inhibiting grasping behaviour.

The raw score is corrected for age and education according to normative reference values.

Digit Span (forward and backward) (Monaco et al., 2013): this test measures verbal short-term memory, in particular the ability to retain and repeat sequences of digits. The examiner reads a sequence of numbers of increasing length and the patient has to repeat the sequence immediately after the presentation. If the patient repeats a sequence correctly, the examiner proceeds with a subsequent longer sequence until the patient makes two consecutive mistakes or fails to repeat a nine-digit sequence correctly. The final score is given by the number of digits of the longest sequence repeated correctly, which varies in length from 3 to 9 digits. The raw score is corrected for age and education according to normative reference values.

Corsi Block Task (forward) (Spinnler and Tognoni, 1987): This is a test that measures the 'span' capacity of visuospatial memory, i.e. the amount of visuospatial information that can be held in short-term memory (STM). The stimulus consists of a 32 cm x 25 cm wooden board on which 9 asymmetrically arranged cubes are glued. The cubes are numbered from the side facing the examiner, not the side facing the patient. The examiner stands in front of the subject and touches the cubes with his index finger in a standard sequence of increasing length (from two to ten cubes). At the end of the demonstration, the examiner asks the subject to reproduce the sequence by touching the cubes in the exact order. If the subject reproduces at least two out of three sequences correctly, the next series is tested. The score is the number of cubes in the longest series for which at least two sequences have been correctly reproduced. The raw score is corrected for age and education according to normative reference values.

Clock Drawing Test (CDT) (Cafarra et al., 2011): is a test that assesses visuoconstructive functions, mental representation, visuospatial orientation, but also planning and symbolic association. The patient is asked to draw the face of a clock, place the numbers correctly and draw the hands to indicate the time '11:10'. The scoring procedure provides for a maximum total score of 15 points, divided into four main categories:

* Contour of the dial (maximum 2 points): evaluation of the shape, closure and proportions of the circle;
* Numbering (maximum 4 points): correctness of the number sequence, positioning, orientation and spacing of the numbers from 1 to 12;
* Hands (maximum 8 points): distinction between the hour and minute hands, correct orientation and congruence with the required time;
* Centre of the watch (maximum 1 point): presence and correct positioning of the centre from which the hands start.

The raw score is corrected for age and education according to the normative reference values.

Symbol Digit Modalities Test (Smith et al., 1968; Amodio et al., 2002): is a test designed to assess cognitive processing speed and working memory. The test consists of a grid containing symbols associated with the numbers 1 to 9. The patient is asked to write down the number corresponding to each symbol and to complete the task as quickly as possible, typically within 90 seconds. During administration, the patient is given the sheet of symbols and must quickly match the number with each symbol. The test can be administered in written form or, if the patient has motor or other difficulties, it can be adapted for oral administration in which the patient verbally states the number corresponding to the symbol. The score is determined by the number of correct answers given by the patient within the time limit, with a score ranging from 0 to 90. The results are compared and corrected with normative values according to age and level of education.

Attention Matrices (Spinnler and Tognoni, 1987): This is a test of selective attention. The test consists of 3 grids, each containing numbers, and the patient has to cross out with a pencil as quickly as possible all the numbers corresponding to those indicated at the top of the matrix. Row A serves as an example. If the subject shows that he/she has understood the task, he/she moves on without further correction to row B, which serves as a warm-up. The subject's performance is counted from line I (line A-B is not counted). The maximum time for each matrix is 45 seconds and is counted from the moment the subject finishes the run-in. The respondent may finish the run-in after the time limit, but only the items correctly crossed out within the time limit will be counted. One point is awarded for each correct item for each of the three matrices presented. The raw score ranges from 0 to 60 and is equal to the sum of the points obtained for the three matrices. The results are compared and corrected with normative values according to age and level of education.

Activities of Daily Living (ADL) (Katz et al., 1963): is a test to assess functional independence in basic activities of daily living. This test is used to measure a person's level of independence in performing essential tasks of daily living. It assesses 6 basic activities:

1. Bathing (washing independently or with partial/full assistance);
2. Dressing (choosing and putting on clothes, fastening buttons, zips);
3. Toileting (getting in and out, using the toilet, toileting);
4. Mobility (getting up and sitting down from bed or chair without assistance);
5. Continence (urinary sphincter and bowel control);
6. Eating (eating alone or with assistance). The total score ranges from 0 to 6 and for each activity the patient receives a binary score: 1 point if the activity is performed independently; 0 points if partial or total assistance is required.

Instrumental Activities of Daily Living (IADL) (Lawton & Brody, 1969): This test assesses a person's ability to perform more complex activities of daily living than ADLs. This test is used to determine whether a patient can perform 8 activities that require planning and the use of cognitive skills:

1. Household and household chores;
2. Taking medication;
3. Getting out of the house;
4. Managing money and household accounts;
5. Preparing meals;
6. Using the telephone or other technology;
7. Using the washing machine;
8. Shopping. The total score ranges from 0 to 8 and for each activity the patient receives a binary score: 1 point if the activity is performed independently; 0 points if partial or total assistance is required.

Neuropsychiatric Inventory (NPI) (Cumming et al., 1994; Binetti et al., 1998): is a questionnaire administered by an expert examiner to the carer. It is a very useful tool for assessing the presence and severity of psychiatric and behavioural disorders in patients with dementia of different aetiologies and their impact on the caregiver's well-being. The questions asked relate to events and changes following cognitive changes. The areas investigated are:

* Delusions;
* Hallucinations;
* Agitation;
* Depression/dysphoria;
* Anxiety;
* Euphoria/exaltation;
* Apathy/indifference;
* Disinhibition;
* Irritability/aggressiveness;
* Motor activity;
* Sleep;
* Appetite and eating disorders. Each behavioural or psychological symptom is rated according to its frequency and severity, and the total score is calculated by combining the two factors for each symptom (frequency × severity), ranging from 0 to 12.

World Health Organisation Quality Of Life Questionnaire-Bref (WHOQOL Group, 1998; De Girolamo et al., 2000): is an abbreviated version of the World Health Organisation Quality Of Live-100 (WHOQOL), a questionnaire developed by the World Health Organisation (WHO) to assess quality of life and subjective well-being in various domains of life. It consists of 26 items, the first two of which measure general quality of life and satisfaction with health. The other 24 items are divided into 4 domains:

1. Physical (pain, energy, sleep, activities of daily living, mobility, medication);
2. Psychological (body image, positive/negative emotions, self-esteem, spirituality);
3. Social (social support, personal relationships, sex life);
4. Environmental (safety, economic resources, leisure, housing, transport, health, information).

Each item is rated on a 5-point Likert scale, with 1 indicating a low quality of life and 5 indicating a high quality of life. To calculate a domain, the average of the scores of the items composing it is calculated. The average scores thus obtained are multiplied by 4 to make them comparable to those of the WHOQOL-100 and then converted to a scale from 0 to 100. Some items are subtracted from 6 because in the WHOQOL-Bref some questions are worded in the opposite way to the meaning of the scale.

Otorhinolaryngology Total time for all tests including complete smell test 40- 60 minutes

1. Sniffin' sticks smell test for threshold (T), detection (D) and identification (I) assessment. Patients will be assessed first by nasal endoscopy and Sniff Test. To ensure objectivity in the analysis, the physician who will perform the Sniffin' checks at the various follow-ups will be blinded to the group to which the patient belongs at the time of the test. Olfactory function will be assessed using the Sniffin' Sticks battery following the standardized TDI (threshold, discrimination, identification) procedure. The Sniffin' Sticks battery consists of pen-like devices filled with odors. Three subtests will be performed to assess orthonasal olfactory function: detection threshold (the lowest concentration at which an odor can be perceived), odor discrimination (the ability to distinguish between odors), and odor identification (the ability to name odors). The odor detection threshold will be identified for each participant using a three-alternative, single-ladder forced-choice procedure with the odor n-butanol. Therefore, participants will be presented with triplets of odorant pens and asked to identify the pen containing n-butanol between two empty distractor pens. In the second test, odor discrimination ability will be assessed using 16 triplets of odorants: within each triplet, two pens will contain the same odorant, while the third pen will contain a different odorant. In a forced-choice procedure, participants will be asked to detect the odd-numbered pen for each triplet. During the odor identification task, participants will be presented with 16 common odorants. Using a multiple-choice format, they will be asked to select which of four odor labels corresponds to each odor presented. Possible scores range from 1 to 16 for the subtest of detection threshold and from 0 to 16 for the other two subtests. The total TDI score is obtained by adding the scores from all three subtests. Normosmia is defined by a TDI score ≥31, hyposmia by a TDI score of 17 to 30.75, and anosmia by a TDI score <17.
2. Tonal and vocal audiometric test
3. Vestibular tests: - nose indices, - Romberg, spontaneous and gaze-evoked NY, Dix-Halpike, Head Shaking Ny,

Radiological investigations

3T brain magnetic resonance with and without contrast, with evaluation of the cortical thickness of the entire brain and of the temporal lobe and evaluation of micro-angiopathy using Fazekas score.

Doppler of the epiaortic vessels of the neck

In case of diagnostic doubt: PET with FdG and Scintifigraphy with dat Scan

ELIGIBILITY:
Inclusion Criteria:

* Patients between 60 and 85 years of age
* in general good health
* the absence of known severe psychiatric disorders
* available to be included in the study and
* to follow the 5-year follow-up.

Exclusion Criteria:

* Obstructive nasal problems
* Previous endoscopic nose + paranasal sinus surgery
* Chronic use of cortisone spray and/or systemic
* Subjects with previous stroke and outcomes
* Subjects with history of stroke in the last 3 years without outcomes
* Head trauma in the last 24 months
* Previous ear surgery
* Patients who have been exposed to chemical agents without protection for work, e.g. carpenters
* previous Covid with outcomes (olfactory, vestibular, auditory and cognitive "brain fog")

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients affected by mild cognitive impairment (MCI), Alzheimer Disease in Early stage, Parkison Disease in early stage
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Impact of hearing loss, vertigo and smell loss on cognition | 5 years
  All these measures are numeric. Vertigo will be yes (1) or no (0), same for hearing loss and smell loss

OTHER OUTCOMES:
Hearing Loss | each year for 5 years
  The hearing capacity will be evaluated by pure tone test
Smell loss | each year for 5 years
  Smell loss will be evaluted by Sniffin' sticks
Vertigo | each year for 5 years
  Walking and standing tests will be performed to evaluate patients stability

CONTACTS AND LOCATIONS:
Locations (1):
- Vanvitelli ENT department, Naples, Campania, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Myrstad C, Engdahl BL, Costafreda SG, Krokstad S, Lin F, Livingston G, Strand BH, Ohre B, Selbaek G. Hearing impairment and risk of dementia in The HUNT Study (HUNT4 70+): a Norwegian cohort study. EClinicalMedicine. 2023 Dec 4;66:102319. doi: 10.1016/j.eclinm.2023.102319. eCollection 2023 Dec. PMID 38192588
- [Result] O'Malley PG. Evolving insights about the impact of sensory deficits in the elderly: comment on "The prevalence of concurrent hearing and vision impairment in the United states" and "Hearing loss and cognitive decline in older adults". JAMA Intern Med. 2013 Feb 25;173(4):299. doi: 10.1001/jamainternmed.2013.3760. No abstract available. PMID 23338615
- [Result] Rong H, Lai X, Jing R, Wang X, Fang H, Mahmoudi E. Association of Sensory Impairments With Cognitive Decline and Depression Among Older Adults in China. JAMA Netw Open. 2020 Sep 1;3(9):e2014186. doi: 10.1001/jamanetworkopen.2020.14186. PMID 32990739
- [Result] Mahmoudi E. Hearing, Vision, or Dual Sensory Impairment and Dementia Risk. JAMA Netw Open. 2021 Mar 1;4(3):e211846. doi: 10.1001/jamanetworkopen.2021.1846. No abstract available. PMID 33739427
- [Result] Liljas AEM, Jones A, Cadar D, Steptoe A, Lassale C. Association of Multisensory Impairment With Quality of Life and Depression in English Older Adults. JAMA Otolaryngol Head Neck Surg. 2020 Mar 1;146(3):278-285. doi: 10.1001/jamaoto.2019.4470. PMID 32027340
- [Result] Stickel AM, Mendoza A, Tarraf W, Kuwayama S, Kaur S, Morlett Paredes A, Daviglus ML, Testai FD, Zeng D, Isasi CR, Baiduc RR, Dinces E, Lee DJ, Gonzalez HM. Hearing Loss and Associated 7-Year Cognitive Outcomes Among Hispanic and Latino Adults. JAMA Otolaryngol Head Neck Surg. 2024 May 1;150(5):385-392. doi: 10.1001/jamaoto.2024.0184. PMID 38512278
- [Result] An YY, Lee ES, Lee SA, Choi JH, Park JM, Lee TK, Kim H, Lee JD. Association of Hearing Loss With Anatomical and Functional Connectivity in Patients With Mild Cognitive Impairment. JAMA Otolaryngol Head Neck Surg. 2023 Jul 1;149(7):571-578. doi: 10.1001/jamaoto.2023.0824. PMID 37166823
- [Result] Lee EY, Eslinger PJ, Du G, Kong L, Lewis MM, Huang X. Olfactory-related cortical atrophy is associated with olfactory dysfunction in Parkinson's disease. Mov Disord. 2014 Aug;29(9):1205-8. doi: 10.1002/mds.25829. Epub 2014 Jan 30. PMID 24482154
- [Result] Kollndorfer K, Jakab A, Mueller CA, Trattnig S, Schopf V. Effects of chronic peripheral olfactory loss on functional brain networks. Neuroscience. 2015 Dec 3;310:589-99. doi: 10.1016/j.neuroscience.2015.09.045. Epub 2015 Sep 28. PMID 26415766
- [Result] Lin FR, Ferrucci L. Hearing loss and falls among older adults in the United States. Arch Intern Med. 2012 Feb 27;172(4):369-71. doi: 10.1001/archinternmed.2011.728. No abstract available. PMID 22371929
- [Result] Vohra V, Simonsick EM, Kamath V, Bandeen-Roche K, Agrawal Y, Rowan NR. Physical Function Trajectories and Mortality in Older Adults With Multisensory Impairment. JAMA Otolaryngol Head Neck Surg. 2024 Mar 1;150(3):217-225. doi: 10.1001/jamaoto.2023.4378. PMID 38236596
- [Result] Di Stadio A, Ralli M, Kaski D. Multisensory Rehabilitation in Older Adults to Improve Longevity and Wellness. JAMA Otolaryngol Head Neck Surg. 2024 Aug 1;150(8):748-749. doi: 10.1001/jamaoto.2024.1695. No abstract available. PMID 38935395